CLINICAL TRIAL: NCT04094740
Title: Effect of Insulin Administered by Needle-free Jet Injection on Blood Glucose Control and Injection Feelings in Patients With Type 1 Diabetes
Brief Title: Effect of Needle-free Jet Injection of Insulin on Glucose Control and Injection Feelings in Type 1 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xia Li, Professor, Department of Endocrinology, Institute of of Metabolism and Endocrinology, Nationa Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JI-EC T1D 2019
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Needle-free Jet Injector (Experimental): Subjects will be instructed to use a needle-free syringe to inject insulin during the study period. The dosage and frequency of insulin are determined by the responsible physician according to the patient's condition.
  Interventions: Device: Jet Injector without A Needle
- Conventional Insulin Pen (No Intervention): Patients allocated to the control group will be instructed to use conventional insulin pens to inject insulin. Except for the syringe, all of them are the same as the experimental group.
- Routine Care (No Intervention): Subjects can receive the education provided by health-care professionals and training in the outpatient department and inpatient departments.

INTERVENTIONS:
Device: Jet Injector without A Needle — Patients in the experimental group will use a needle - free jet injector to inject insulin, which delivers insulin at a high velocity into subcutaneous tissue and dispenses insulin over a larger area than a syringe.
  Arms: Needle-free Jet Injector

SUMMARY:
People with type 1 diabetes need long-term insulin injections. However, needles may cause discomfort or provoke anxiety if the patient has needle phobia, factors that contribute to poor compliance with insulin, especially in younger patients. Use of needle-free technology has been proposed as a strategy to mitigate these problems. There have been few studies on the efficacy of needle-free syringes for patients with type 1 diabetes. To determine the efficacy of needle-free injection of insulin in its patient population, people with type 1 diabetes, we conduct a pilot study to assess glycemic control and injection experience of patients. For the comparator device, we used an insulin pen. The primary objective is to explore whether needle-free syringes are more beneficial to control blood glucose than insulin pens of type 1 diabetes, which the blood sugar fluctuates significantly. The secondary objective is to evaluate the experience and safety of insulin administration by the needle-free injection.

DETAILED DESCRIPTION:
This is a single-center, prospective, 1:1 parallel-group, randomized controlled trial. The intervention will last for 12 weeks. The laboratory staff who tests the HbA1c level, the outcome assessor who collects the blood glucose data and injection experience include the measurement of perceived pain, skin condition at the injection site, and device preference in participants, and the statisticians will be blinded to the treatment allocation.

After informed consent is obtained, the participants can attend an initial study visit to determine eligibility for the trial. We propose to enroll 60 patients with type 1 diabetes (T1DM), participants are randomized into two groups, 30 in the needle-free jet injection group and 30 in the pen injection group. Sample size estimation is based on hypothesized changes in the primary outcome pre-prandial glucose in the morning. Participants are randomized using a computer-generated list.

In order to ensure high quality data, two staff are responsible for the input of original data into the database to check and confirm the accuracy. When the data entered by two people are inconsistent, the auxiliary staff decides which data to use.

Data analysis will be conducted under the intention-to-treat principle by including all the randomized patients in the data analysis. Missing data will be filled in with multiple imputation method. Any substantial difference in baseline characteristics will be adjusted with mixed-model regression analysis. Sensitivity analysis will be conducted by using per-protocol data by excluding those patients who drop out of the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Type 1 Diabetes according to the 1999 World Health Organization report
* Insulin dependence from disease onset
* Older than 12
* The patient's blood glucose is stable after the washout period (insulin dose is less than 30% compared with the last adjustment).

Exclusion Criteria:

* Recent unstable angina, myocardial infarction, or severe cardiac failure, blood pressure ≥180/100mm Hg, activities of hepatic transaminases >2.5 times the upper limit of normal and estimated glomerular filtration rate <30mL/min/1.73m2
* Being pregnant
* Serious mental problems
* Abuse of alcohol or narcotics
* Use of systemic glucocorticoids
* Have any other condition or disease that may hamper from compliance with the protocol or complication of the trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Continuous Glucose Monitoring(CGM) | from baseline to week 4, 12
  CGM reflects the blood glucose fluctuations in the past 2-3 days.
changes in serum hemoglobin A1c level | from baseline to week 12
  A1c reflects the average blood glucose level in the past 2-3 months.

SECONDARY OUTCOMES:
Visual Analog Scale | From baseline to every 2 weeks
  Visual Analog Scale is used to assess perceived pain in each injection. Participants will complete a visual analog scale in which perceived pain is scored from 0 (no pain) to 10 (worst pain ever).
Insulin Treatment Satisfaction Questionnaire | from baseline to week 2，4，12
  Insulin Treatment Satisfaction Questionnaire (ITSQ) is used to assess the diabetes insulin treatment satisfaction. This scale contains 5-factor, 22-item instrument assessing regimen inconvenience, lifestyle flexibility, glycemic control, hypoglycemic control, and satisfaction with the insulin delivery device. Participants evaluate it based on their treatment experience over the past 4 weeks. Each item is divided into seven grades (1-7 points), and the total score of the scale is the mean score of the five dimensions. Higher score reflects better the satisfaction.
Insulin Treatment Attitude Scale | from baseline to week 2，4，12
  Insulin Treatment Attitude Scale (ITAS) is to assess the attitude of diabetes towards insulin treatment. This scale contains 3 aspects with a total of 20 items, Using the Liket5 scoring method, from strongly disagree (1 point) to strongly agree (5 points), the total score of more than 60 points is considered as the presence of psychological insulin resistance.
Insulin Treatment Adherence Questionnaire | from baseline to week 2，4，12
  Insulin treatment adherence questionnaire (ITAQ) is to assess the diabetes insulin treatment compliance. This scale contains five aspects with a total of 22 items: Medications, diet, exercise, self-monitoring of blood sugar, regular review. Items are graded on a regular basis (1 point), occasionally (2 points), and never (3 points), the total score of more than 44 points is considered as better the compliance.
Adjusted Diabetes Quality of Life Measure (A-DQOL) | from baseline to week 2，4，12
  Adjusted-Diabetes Quality of Life Measure (DQOL) is to assess the quality of life of diabetic patients. This scale contains four aspects with a total of 46 items: satisfaction degree, influence degree, worry degreeⅠand worry degreeⅡ.
Skin condition at the injection site | every 2 weeks from baseline to week 12
  The staff detects the skin condition by the B-mode ultrasound machine to assess whether there is fatty hyperplasia, skin depression, etc.
Fasting blood glucose | From baseline to every 2 weeks
  the blood sugar level after fasting for eight hours
Systolic blood pressure | from baseline to week 4，12
  Systolic blood pressure
Diastolic blood pressure | from baseline to week 4，12
  Diastolic blood pressure
Height in meters | from baseline to week 4，12
  Height in meters will be measured
Weight in kilograms | from baseline to week 4，12
  Weight in kilograms will be measured.
Total daily dose of insulin | every 2 weeks from baseline to week 12
  Contains all insulin doses for the day
Adverse events | every 2 weeks from baseline to week 12
  Safety-related outcomes including hypoglycemic events, hospitalization, and emergency room visits will be collected at each follow-up time point including the weekly telephone interview.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Li, MD/PHD, Principal Investigator — Central South University

IPD SHARING:
Plan to Share IPD: No